CLINICAL TRIAL: NCT01965184
Title: Using CBT to Examine Circuitry of Frustrative Non-reward in Aggressive Children
Brief Title: Cognitive-Behavioral Therapy for Disruptive Behavior in Children and Adolescents
Acronym: RDoC-CBT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0102012121-C; R01MH101514 (NIH)
Record Dates: First submitted 2013-10-14; First posted 2013-10-18 (Estimated); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Disruptive Behavior; Aggression; Anger; Irritability; Noncompliance
Keywords: child; cognitive behavioral therapy; CBT; aggression; disruptive behavior; treatment; frustrative non-reward; irritability
MeSH Terms: conditions — Problem Behavior; Aggression; Patient Compliance | interventions — Cognitive Behavioral Therapy; mycophenolic adenine dinucleotide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cognitive-Behavioral Therapy for Anger and Aggressive Behavior (Experimental): CBT is a behavioral intervention that consists of 12 weekly sessions. During CBT children are taught various skills for coping with frustration and parents are taught various strategies for managing situations that can be anger provoking for their child.
  Interventions: Behavioral: Cognitive-Behavioral Therapy for Anger and Aggression
- Supportive Psychotherapy (SPT) (Active Comparator): SPT consists of 12 sessions that are focused on discussing peer relationships and family functioning with a goal of enhancing subjective well-being
  Interventions: Behavioral: Supportive Psychotherapy (SPT)

INTERVENTIONS:
Behavioral: Cognitive-Behavioral Therapy for Anger and Aggression
  Arms: Cognitive-Behavioral Therapy for Anger and Aggressive Behavior
Behavioral: Supportive Psychotherapy (SPT)
  Arms: Supportive Psychotherapy (SPT)

SUMMARY:
This is a randomized controlled study of cognitive-behavioral therapy (CBT) for disruptive behavior such as irritability, anger and aggression in children and adolescents. CBT will be compared to Supportive Psychotherapy (SPT) and participants of this study will be randomly assigned (like the flip of a coin) to receive CBT or SPT. Participants will be also asked to complete functional magnetic resonance imaging (fMRI) and electrophysiological (EEG) tasks (recordings/images of brain activity) before and after treatment.

DETAILED DESCRIPTION:
Cognitive-behavioral therapy (CBT) is a behavioral intervention that consists of 12 weekly sessions. During CBT children are taught various skills for coping with frustration and parents are taught various strategies for managing situations that can be anger provoking for their child. This study is conducted to examine whether reduction of behavioral problems including anger outbursts, irritability, aggression and noncompliance after CBT may be paralleled by changes in areas of the brain responsible for emotion regulation and social perception.

ELIGIBILITY:
Inclusion Criteria:

1. Boys and girls, 8 to 16 years of age.
2. T-Score > 65 on the parent-rated Aggressive Behavior Scale of the Child Behavior Checklist (CBCL).
3. Unmedicated or on stable medication for aggression, ADHD, anxiety, or depression for at least 6 weeks, with no planned changes for duration of study.
4. Children can speak English sufficiently enough to participate in CBT and study assessments.
5. Children should have 1) no metal medical implants, 2) a body weight of less than 250 lbs. and 3) no claustrophobia. [These are necessitated by the safety requirements of the fMRI.]
6. Children should be able to meet fMRI data quality requirements at baseline [to enable pre- to post-treatment comparison.]
7. Families can commute to the Yale Child Study Center in New Haven, CT for weekly visits.

Exclusion Criteria:

1. IQ below 85.
2. Children across various DSM diagnoses will be eligible for participation. However, significant levels of psychopathology that require immediate clinical attention such as severe depression or psychosis will be exclusionary because it will require alternative treatments.
3. Significant medical condition such as heart disease, hypertension, liver or renal failure, pulmonary disease, seizure disorder, brain injury based on medical history which can interfere with participation in the study.
4. Concurrent psychotherapy can continue, but CBT for aggression is exclusionary. Subjects will be asked not to initiate any new child psychotherapy during the study.

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 101 (Actual)
Dates: Start 2013-11-14 (Actual); Primary Completion 2018-08-03 (Actual); Study Completion 2018-11-03 (Actual)

PRIMARY OUTCOMES:
Modified Overt Aggression Scale | basline (week 0)
  Modified Overt Aggression Scale is a 16-item scale that reflects the frequency and severity of incidents of aggressive behavior. Scores can range from 0 (minimum) to 300 (maximum) with higher scores reflecting worse outcome.
Modified Overt Aggression Scale | midpoint (week 6)
  Modified Overt Aggression Scale is a 16-item scale that reflects the frequency and severity of incidents of aggressive behavior. Scores can range from 0 (minimum) to 300 (maximum) with higher scores reflecting worse outcome.
Modified Overt Aggression Scale | endpoint (week 12)
  Modified Overt Aggression Scale is a 16-item scale that reflects the frequency and severity of incidents of aggressive behavior. Scores can range from 0 (minimum) to 300 (maximum) with higher scores reflecting worse outcome.
Modified Overt Aggression Scale | follow up (3 months)
  Modified Overt Aggression Scale is a 16-item scale that reflects the frequency and severity of incidents of aggressive behavior. Scores can range from 0 (minimum) to 300 (maximum) with higher scores reflecting worse outcome.
The Clinical Global Impression - Improvement Score | basline (week 0)
  The Clinical Global Impression - Improvement Score assigned by an independent evaluator (IE) who will be blind to treatment assignment is the categorical primary outcome measure of aggressive behavior. The CGI-I reflects the IE's assessment of overall change from baseline rated on a scale from 1 to 7 where 1 is very much improved, 2 is much improved, 3 is minimally improved, 4 is no change, 5 is minimally worse, 6 is much worth, and 7 is very much worse. Higher scores reflect worse outcome. By convention, ratings of very much improved (1) or much improved (2) define positive response; all other scores are classified as a negative response.
The Clinical Global Impression - Improvement Score | midpoint (week 6)
  The Clinical Global Impression - Improvement Score assigned by an independent evaluator (IE) who will be blind to treatment assignment is the categorical primary outcome measure of aggressive behavior. The CGI-I reflects the IE's assessment of overall change from baseline rated on a scale from 1 to 7 where 1 is very much improved, 2 is much improved, 3 is minimally improved, 4 is no change, 5 is minimally worse, 6 is much worth, and 7 is very much worse. Higher scores reflect worse outcome. By convention, ratings of very much improved (1) or much improved (2) define positive response; all other scores are classified as a negative response.
The Clinical Global Impression - Improvement Score | endpoint (week 12)
  The Clinical Global Impression - Improvement Score assigned by an independent evaluator (IE) who will be blind to treatment assignment is the categorical primary outcome measure of aggressive behavior. The CGI-I reflects the IE's assessment of overall change from baseline rated on a scale from 1 to 7 where 1 is very much improved, 2 is much improved, 3 is minimally improved, 4 is no change, 5 is minimally worse, 6 is much worth, and 7 is very much worse. Higher scores reflect worse outcome. By convention, ratings of very much improved (1) or much improved (2) define positive response; all other scores are classified as a negative response.
The Clinical Global Impression - Improvement Score | follow up (3 months)
  The Clinical Global Impression - Improvement Score assigned by an independent evaluator (IE) who will be blind to treatment assignment is the categorical primary outcome measure of aggressive behavior. The CGI-I reflects the IE's assessment of overall change from baseline rated on a scale from 1 to 7 where 1 is very much improved, 2 is much improved, 3 is minimally improved, 4 is no change, 5 is minimally worse, 6 is much worth, and 7 is very much worse. Higher scores reflect worse outcome. By convention, ratings of very much improved (1) or much improved (2) define positive response; all other scores are classified as a negative response.

SECONDARY OUTCOMES:
The Child Behavior Checklist | basline (week 0)
  The Child Behavior Checklist is a parent rating of child psychopathology that has two factor-analytically derived scales of disruptive behavior. Child Behavior Checklist Aggressive Behavior Scale consists of 18 items, rated as 0, 1 or 2, with a scale raw score range from 0 (minimum) to 36 (maximum) with higher scores reflecting worse outcome. Raw scores are also converted to T-scores with possible range from 0 to 100 with higher scores reflecting worse outcomes and T-scores of 65 and higher reflecting clinically significant range.
The Child Behavior Checklist | midpoint (week 6)
  The Child Behavior Checklist is a parent rating of child psychopathology that has two factor-analytically derived scales of disruptive behavior. Child Behavior Checklist Aggressive Behavior Scale consists of 18 items, rated as 0, 1 or 2, with a scale raw score range from 0 (minimum) to 36 (maximum) with higher scores reflecting worse outcome. Raw scores are also converted to T-scores with possible range from 0 to 100 with higher scores reflecting worse outcomes and T-scores of 65 and higher reflecting clinically significant range.
The Child Behavior Checklist | endpoint (week 12)
  The Child Behavior Checklist is a parent rating of child psychopathology that has two factor-analytically derived scales of disruptive behavior. Child Behavior Checklist Aggressive Behavior Scale consists of 18 items, rated as 0, 1 or 2, with a scale raw score range from 0 (minimum) to 36 (maximum) with higher scores reflecting worse outcome. Raw scores are also converted to T-scores with possible range from 0 to 100 with higher scores reflecting worse outcomes and T-scores of 65 and higher reflecting clinically significant range.
The Child Behavior Checklist | follow up (3 months)
  The Child Behavior Checklist is a parent rating of child psychopathology that has two factor-analytically derived scales of disruptive behavior. Child Behavior Checklist Aggressive Behavior Scale consists of 18 items, rated as 0, 1 or 2, with a scale raw score range from 0 (minimum) to 36 (maximum) with higher scores reflecting worse outcome. Raw scores are also converted to T-scores with possible range from 0 to 100 with higher scores reflecting worse outcomes and T-scores of 65 and higher reflecting clinically significant range.

OTHER OUTCOMES:
functional magnetic resonance imaging (fMRI) | baseline (week 0)
  fMRI scanning with tasks of emotion regulation and social perception
Electroencephalography (EEG) | baseline (week 0)
  EEG recordings will be collected as participants perform tasks of emotion regulation and social perception
functional magnetic resonance imaging (fMRI) | endpoint (week 12)
  fMRI scanning with tasks of emotion regulation and social perception
Electroencephalography (EEG) | endpoint (week 12)
  EEG recordings will be collected as participants perform tasks of emotion regulation and social perception

CONTACTS AND LOCATIONS:
Overall Officials: Denis G. Sukhodolsky, Ph.D., Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

REFERENCES:
- [Background] Sukhodolsky, D. G. & Scahill, L. (2012). Cognitive-behavioral therapy for anger and aggression in children. New York: Guilford Press.
- [Background] Sukhodolsky DG, Vitulano LA, Carroll DH, McGuire J, Leckman JF, Scahill L. Randomized trial of anger control training for adolescents with Tourette's syndrome and disruptive behavior. J Am Acad Child Adolesc Psychiatry. 2009 Apr;48(4):413-421. doi: 10.1097/CHI.0b013e3181985050. PMID 19242384
- [Background] Perlman SB, Pelphrey KA. Developing connections for affective regulation: age-related changes in emotional brain connectivity. J Exp Child Psychol. 2011 Mar;108(3):607-20. doi: 10.1016/j.jecp.2010.08.006. Epub 2010 Oct 23. PMID 20971474